CLINICAL TRIAL: NCT02901561
Title: Comparison Between 2 Different Doses of Vaginal Misoprostol Before Intrauterine Device Insertion in Parous Women
Brief Title: Comparison Between 2 Doses of Misoprostol Before Intrauterine Device
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MISO
Record Dates: First submitted 2016-09-10; First posted 2016-09-15 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Pain Relief

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol 200 (Experimental): misoprostol 200 microgram placed into the vagina 3 hours prior to having the intrauterine device inserted
  Interventions: Drug: misoprostol 200
- misoprostol 400 (Active Comparator): misoprostol 400 microgram placed into the vagina 3 hours prior to having the intrauterine device inserted
  Interventions: Drug: misoprostol 400

INTERVENTIONS:
Drug: misoprostol 200
  Arms: misoprostol 200
Drug: misoprostol 400
  Arms: misoprostol 400

SUMMARY:
The purpose of the investigators' study was to evaluate whether misoprostol will improve pain scores .

DETAILED DESCRIPTION:
an intrauterine device can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the intrauterine device insertion tube, and removing the tube; and placement of the device in the uterus.

ELIGIBILITY:
Inclusion Criteria:

* • Women not taken analgesics or anxiolytics in the 24 hours prior insertion

  * Women who will accept to participate in the study

Exclusion Criteria:

* Any contraindication to IUD placement

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mean pain score during intrauterine device insertion | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes